# PMCF Study on PEEK Suture Anchors for Hip Indications

Protocol Number: 2018.14.SMD.PEEK.RET.HIP

Protocol Version: Version 2.0
Date: 03 April 19

Study Product Names: PEEK Hip Suture Anchors

Bioraptor Knotless Suture Anchor SpeedLock Hip Suture Anchor

Sponsor: Smith & Nephew Orthopaedics

7135 Goodlett Farms Parkway

Cordova, TN 38016

#### ****

| Study Protocol—Device | smith&nephew |
|-------------------------------------------|----------------------------------|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| • | Version: 2.0, 03 April 2019 |
| Indications | |

# 1. SIGNATURES

# 1.1 PROTOCOL SIGNATURE PAGE

This page will be returned to Smith & Nephew Inc. and a copy retained at the investigational site.

I have read the attached protocol entitled "PMCF Study on PEEK Suture Anchors for Hip Indications", version 2.0, dated 03April2019, and agree to abide by all provisions set forth herein.

I agree to comply with the Investigator's Obligations stipulated in Section 26.1 of the protocol, I agree to ensure that the confidential information contained in this document will not be used for any purpose other than the conduct of the described clinical investigation without the prior written consent of Smith & Nephew, Inc.

| Role | Name | Signature* | Date Signed* (DD-MMM-YYYY) |
|------------------------|------|------------|----------------------------|
| Principal Investigator | | | |

### ****

| Study Protocol—Device | > smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| , | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

- 2. REVISION HISTORY, OWNERSHIP, AND APPROVALS:
- **2.1 REVISION HISTORY**

[Intentionally left blank]

# ****

| Study Protocol—Device | > smith&nephew |
|---|---|
| DMCF Study on DEFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

| Version | Page | Item | Original | | | New | | | | Reason | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1.0 | N/A | N/A | Initial Protocol | | | Revision 2.0 | | | | N/A | |
| 2.0 | 2 | Protocol<br>Signature Page | 1.0<br>12Sep18 | | | 2.0<br>03April19 | | | | Administrative | |
| 2.0 | ဇ | Revision<br>History | Initial | | | Protocol Amendment 2 | ndment 2 | | | Administrative | |
| 2.0 | 19 | Signatures | Sponsor Signatures | ıtures | | Removed dup | Removed duplicate sponsor signature lines | nature lines | | Administrative | |
| 2.0 | 20, 32 | Part Numbers | N/A | | | Added: Part n | Added: Part numbers as of September 2018 | tember 2018 | | Administrative | |
| 2.0 | 20 | Min/Max | Minimum, n=40 | 01 | | Minimum num | Minimum number of subjects, n=40 | 1=40 | | Administrative/Clarification | Ę |
| | | | Maximum, n=80 | 80 | | Maximum nur | Maximum number of subjects, n=240 | n=240 | | | |
| 2.0 | 20 | Enrollment | N/A | | | Enrollment distribution: | tribution: | | | Rationale for enrollment | |
| | | Distribution | | | | Up to three sil<br>anchor config<br>will be enrolle | Up to three sites will enroll a maximum of 40 subjects per<br>anchor configuration; therefore, no more than 120 subjects<br>will be enrolled for any anchor type. | aximum of 40 sub<br>no more than 12º<br>ype. | o subjects | distribution among sites and between anchors. | |
| 2.0 | 21 | Sample Size | PEEK | Minimum | Maximum | PEEK | Minimum | Maximum | Maximum | Administrative/Clarification | ٦ |
| | i | | Anchor | | | Anchor | Number of | Number of | Number | | |
| | | | Bioraptor<br>Knotless | 20 | 40 | | Subjects/Site | Subjects/Site | of<br>Subjects | | |
| | | | Suture<br>Anchor | | | | | | | | |

| Study Protocol—Device | * smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | |

| Reason | | | | | | | | Clarification | | | | | | Clarification | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | for the<br>Study | 120 | subjects | | 120 | subjects | 240<br>subjects | ļ — | | time of | | provider | ນ່ | | onal drug, | ated with | s prior to | | |
| | | 40 subjects | per site | | 40 subjects | per site | 80 subjects | dergone shoulder | ý | and older at the | | ad a visit to their p | IIIs post-operaliv | months post-ope | nother investigati | ly or has been tre | uct within 30 day | | |
| | | 20 subjects | per site | | 20 subjects | per site | 40 subjects | Subjects who have undergone shoulder joint repair | using the study devices. | Subjects aged 18 years and older at the time of | ery. | Subjects must have had a visit to their provider | between 3 and 13 monins post-operative. | Subjects who are < 12 months post-operative. | Subject is entered in another investigational drug, | biologic, or device study or has been treated with | an investigational product within 30 days prior to | ery. | |
| New | | Bioraptor | Knotless | Suture<br>Anchor | SpeedLock | Нiр | Total | 1. Subje | guisn | 2. Subje | surgery. | 3. Subj | Delw | 1. Subje | 2. Subje | goloid | an in | surgery. | |
| | 40 | | | | | | | ve undergone | air using the | | years and | ime of surgery. | | < 12 months | | d in another | ug, biologic, | r has been | ivestigational |
| | k 20 | | | | | | | Subjects who have undergone | shoulder joint repair using the | ıdy devices. | | older at the time | | Subjects who are < 12 months | post-operative. | Subject is entered in another | investigational drug, biologic, | or device study or has been | treated with an investigational |
| Original | SpeedLock<br>Hip | | | | | | | 1. Su | - S | otc | 2. Su | olo<br> | | 1. Su | Ö. | 2. Su | inv | oľ | tre |
| Item | | | | | | | | Inclusion | Criteria | | | | | Exclusion | Criteria | | | | |
| Version | | | | | | | | 2.0 | | | | | | 2.0 | | | | | |

| Study Protocol—Device | smith&nephew |
|-------------------------------------------|----------------------------------|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| | Version: 2.0, 03 April 2019 |
| Indications | |

| Reason | | Clarification | Clarification | Clarification | Clarification | Administrative | Administrative | Administrative |
|---|---|---|---|---|---|---|---|---|
| | Subject had off-label use of the PEEK suture anchorduring surgery. | months post-operative based | Clinical success rate (%) at 12 months post-operative based on standard of care. | ed by IRB | mpleted at 6 months if the nth visit. | | | IFU |
| New | 3. Subject had off-label during surgery. | Clinical success rate (%) at 6 months post-operative based on standard of care. | Clinical success rate (%) at 12 on standard of care. | NA if waiver of consent granted by IRB | <sup>2</sup> End of Study CRF can be completed at 6 months if the subject did not have a 12-month visit. | Removed. Not applicable. | | PEEK Suture Anchor |
| | product within 30 days prior to surgery. | ite (%) at 6 months | ite (%) at 12 months | NA if waiver of consent approved by IRB | | | | IFU |
| Original | product wit<br>to surgery. | Clinical success rate (post-operative. | Clinical success rate (post-operative. | NA if waiver of cor<br>IRB | NA<br>A | BMI<br>PHI<br>PROs | | PEEK Suture<br>Anchor |
| Item | | Primary<br>Endpoint | Secondary<br>Endpoint | SOE/ICF | SOE/Footnote | List of<br>Abbreviations | Minor<br>formatting<br>corrections | IFUs |
| Page | | 21, 37 | 21, 37 | 23 | 23 | 27 | Throughout | 30 |
| Version | | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 | 2.0 |

| Study Protocol—Device | * smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Page: 7</b> of <b>63</b> |

| Reason | | | | Clarification | Clarification | | | Clarification | | | | | | Clarification | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 10600479 2/17, Rev E<br>P/N 62513 March 2017. | Rev B | | Instructions for Use document numbers have been provided as a reference but may not have been the version used at the time of surgery. | | their surgical procedure with the investigational device, i.e. | зу. | Subjects who have undergone shoulder joint repair | rices. | Subjects aged 18 years and older at the time of | | Subjects must have had a visit to their provider | between 3 and 15 months post-operative. | Subjects who are < 12 months post-operative. | Subject is entered in another investigational drug, | biologic, or device study or has been treated with | |
| New | Bioraptor Knotless Suture Anchor SpeedLock Hip Suture | Anchor | | Instructions for Use documer as a reference but may not he the time of surgery. | Enrollment will be in sequent | their surgical procedure with | time of surgery to present day. | 1. Subjects who have | using the study devices. | 2. Subjects aged 18 ye | surgery. | 3. Subjects must have | between 3 and 15 n | 1. Subjects who are < | 2. Subject is entered in | biologic, or device s | |
| | 10600479 2/17,<br>Rev E | P/N 62513 | March 2017, Rev<br>B | Ą | sequential order | of their surgical | investigational<br>o latest | Subjects who have undergone | shoulder joint repair using the | ses. | | time of surgery. | | Subjects who are < 12 months | ıtive. | Subject is entered in another | investigational drug, biologic, |
| Original | Bioraptor<br>Knotless Suture<br>Anchor | SpeedLock | | A/N | Enrollment will be in sequential order | based on the date of their surgical | procedure with the investigational device, i.e. earliest to latest. | 1. Subjects w | shoulder jo | study devices. | 2. Subjects a | older at the | | 1. Subjects w | post-operative. | 2. Subject is | investigatic |
| Item | | | | ΙFU | Subject | Population | | Inclusion | Criteria | | | | | Exclusion | Criteria | | |
| Page | | | | 30 | 33 | | | 33 | | | | | | 34 | | | |
| Version | | | | 2.0 | 2.0 | | | 2.0 | | | | | | 2.0 | | | |

| Study Protocol—Device | > smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b></b> |

| Reason | | Removed, as it is not applicable to this study. | Clarification |
|---|---|---|---|
| New | an investigational product within 30 days prior to surgery. 3. Subject had off-label use of the PEEK suture anchor during surgery. | N/A | This is a retrospective, open-label, multicenter study to collect clinical data that will evaluate post-market safety and performance of the PEEK suture anchors in the hip. A minimum of 40 subjects and a maximum of 240 subjects in the United States who underwent surgery in the hip using the Smith & Nephew PEEK suture anchors are planned to be enrolled into the study after the fulfilment of all inclusion and exclusion criteria. Up to three sites will enroll a minimum of 20 subjects and a maximum of 40 subjects per anchor |
| Original | or device study or has been<br>treated with an investigational<br>product within 30 days prior<br>to surgery. | A subject will be considered lost to follow-up if he/she did not return for follow-up per the study doctor's standard of care. | This is a retrospective, open-label, multicenter study to collect clinical data that will evaluate post-market safety and performance of the PEEK suture anchors in the hip. A minimum of 40 subjects and maximum of 80 subjects in the United States who underwent surgery in the hip using the Smith & Nephew PEEK anchor sutures are planned to be enrolled into the study |
| Item | | LTFU | Study Design |
| Version | | 2.0 | 2.0 |

| Study Protocol—Device | > smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Page: 9</b> of <b>63</b> |

| Reason | | Clarification | Clarification |
|---|---|---|---|
| New | configuration; therefore, not more than 120 subjects will be enrolled for any anchor type. | The secondary endpoint will be clinical success rate (%) at 12 months post-operative based on standard of care. Clinical success has previously been defined. It is expected that per physician's standard of care, 12-month clinical data may not be available for all subjects. | Any concomitant medications associated with an AE, SAE or SADE will be recorded. Concomitant medications will be recorded from the time of surgery through 12 months. If the subject's final visit occurred at 6 months, concomitant medications will be collect through 6 months. |
| Original | after the fulfillment of all inclusion and exclusion criteria. It is also planned that each investigational site would enroll a minimum of 6 subjects. | The secondary endpoint will be clinical success rate (%) at 12 months postoperative based on standard of care. Clinical success has previously been defined. | Any concomitant medications associated with an AE, SAE or SADE will be recorded. |
| Item | | Secondary Endpoint | Concomitant<br>Medications<br>and Therapies |
| Version | | 2.0 | 2.0 |

| Study Protocol—Device | > smith&nephew |
|-------------------------------------------|----------------------------------|
| DMCF Study on PEFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | |

| Reason | Clarification | | | | | Clarification | | | Clarification | | Clarification | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| New | Smith & Nephew's Global Biostatistics group or designee will conduct the statistical analysis for this study. Unless | otherwise stated, all significance tests will be two-sided, | performed at the 5% significance level. | | | Resulting p-values will be provided and 95% two-sided | confidence intervals will be generated where appropriate. | | A listing of concomitant medications will be provided by | subject. | The derivation of surgeon reported outcomes used in | summarizing this data for the study will be described in the | SAP and will be summarized as appropriate using descriptive | |
| Original | Smith & Nephew's Global Biostatistics<br>group will conduct the statistical | analysis for this study. Unless | otherwise stated, all significance tests | will be two-sided, performed at the 5% | significance level. | Resulting p-values will be quoted and | 95% two-sided confidence intervals | will be generated where appropriate. | A listing of concomitant medications | will be provided by subject for AEs, | The derivation of surgeon reported | outcomes used in summarizing this | data for the study will be described in | the SAP and will be summarized as |
| Item | General | | | | | General | | | Safety Analysis | | Other Endpoint | Analysis | | |
| Page | 39 | | | | | 39 | | | 41 | | 42 | | | |
| Version | 2.0 | | | | | 2.0 | | | 2.0 | | 2.0 | | | |

| Study Protocol—Device | % smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Page: 11</b> of <b>63</b> |

| Version | Page | Item | Original | New | Reason |
|---|---|---|---|---|---|
| | | | appropriate using descriptive summary | summary characteristics for continuous or categorical | |
| | | | characteristics for continuous or | endpoints at 6 months and 12 months. | |
| | | | categorical endpoints. Differences from | | |
| | | | screening/baseline to 6 months and 12 | | |
| | | | months will be similarly summarized | | |
| | | | and/or compared. | | |
| 2.0 | 42 | | With an assumption of a 91% clinical | With an assumption of a 91% clinical success rate to be | Clarification |
| | | Sample Size | success rate to be obtained in each of | obtained in each of the PEEK anchor sutures and a | |
| | | JUSIIIICAIION | the PEEK anchor sutures and a | corresponding 95% CI between 80% and 100%, enrolling | |
| | | | corresponding 95% CI between 80% | between 20 and 120 subjects for each PEEK anchor suture's | |
| | | | and 100%, enrolling between 20 and | precision analysis will provide between 15.2% to 95% | |
| | | | 40 subjects for each PEEK anchor | probability. Thus, an overall minimum of 40 and maximum of | |
| | | | suture's precision analysis would | 240 subjects who had previously undergone surgery of the | |
| | | | provide between 15.2% to 71% | hip using PEEK anchor sutures will be enrolled into the study. | |
| | | | probability. Thus, an overall minimum | Additionally, a minimum of 20 subjects will be enrolled at any | |
| | | | of 40 and maximum of 80 subjects | investigational site. | |
| | | | who had previously undergone surgery | | |

| Study Protocol—Device | smith&nephew |
|---|---|
| DMCE Study on DEEK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | |

| Reason | | | Clarification implemented as it is applicable for a retrospective study. |
|---|---|---|---|
| New | | All adverse events will be captured from the time of surgery through the 12 month follow-up visit. | AE of any kind and DevD will be recorded in the applicable CRF and source notes. The Investigator will evaluate all AE for relationship to the device and procedure, if applicable, seriousness, and severity. ADE, SAE, and DevD will be entered into the CRF and reported to the Sponsor within 24 hours of the investigator being informed about the event (Figure 1). Applicable to the retrospective study design, 24 hour reporting begins at the time the Investigator was informed of the event under the auspice of the clinical study. |
| Original | of the hip using PEEK anchor sutures would be enrolled into the study. Additionally, a minimum of 6 subjects would be enrolled at any investigational site. | All adverse events will be captured. | AE of any kind and DevD will be recorded in the applicable CRF and source notes. The Investigator will evaluate all AE for relationship to the device and procedure, if applicable, seriousness, and severity. ADE, SAE, and DevD will be entered into the CRF and reported to the Sponsor within 24 hours of the investigator being |
| Item | | AE Definitions | Reporting<br>Procedures |
| Version | | 2.0 | 2.0 |

| Study Protocol—Device | * smith&nephew |
|---|---|
| DMCF Study on DEFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Page: 13</b> of <b>63</b> |

| Reason | edure related | able and | able, the | to S&N unless | ot be | | | | | | | | Clarification implemented | as it is applicable for a | refrospective study | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| New | For ADE and DevD, details of the product/procedure related | to the event will be included and where applicable and | available, pictures taken of the device. If available, the | deficient product should be retained for return to S&N unless | it is contaminated (e.g. used dressings must not be | retained). | | | | | | | Removed | | | |
| Original | informed about the event (Figure 1). | For ADE and DevD, details of the | product/procedure related to the event | will be included and where applicable, | pictures taken of the device. The | deficient product should be retained for | return to S&N unless it is contaminated | (e.g. used dressings must not be | retained). <del>Updates to submitted</del> | information will be recorded in the CRF | within 24 hours of the information | being available to the investigator. | For subjects who are experiencing | ongoing unresolved AE at the time of | their study completion or early | discontinuation from the study, it is |
| Item | | | | | | | | | | | | | Follow-up of | Subjects with | Adverse Events | |
| Page | | | | | | | | | | | | | N/A | | | |
| Version | | | | | | | | | | | | | 2.0 | | | |

| Study Protocol—Device | >/ smith&nephew |
|---|---|
| DMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | |

| Reason | | | | | | | | | Clarification implemented | as it is applicable for a | reirospective study | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| New | | | | | | | | | Removed | | | | | | | | |
| Original | schedule an appropriate follow-up visit | in order to determine the outcome of | the event. | Any additional data must be | documented and available to the | Sponsor who will determine whether | the data need to be documented within | the CRF/Clinical Study Report. | Adverse events which are related to a | study procedure or S&N IP and are | ongoing at end of subject's | participation: The event should be | followed until it is either resolved or | until the event has become chronic and | is not expected to further improve | based on Investigator's review of the | event. |
| Item | | | | | | | | | Ongoing | Adverse Events | at study<br>Discontinuation | | | | | | |
| Page | | | | | | | | | N/A | | | | | | | | |
| Version | | | | | | | | | 2.0 | | | | | | | | |

| Study Protocol—Device | >\ smith&nephew |
|-------------------------------------------|----------------------------------|
| PMCF Study on PFEK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | |

| Reason | | | | | | | | | | | Clarification- Financial | disclosures is not | applicable. | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| New | | | | | | | | | | | Removed | | | | | |
| Original | Adverse events which are not related | to a study procedure or S&N IP and are | ongoing at end of subject's | participation should be followed for 30 | days after discontinuation or if the AE is | resolved, whichever is sooner. | At the time of data analysis (e.g. | interim or final), an evaluation of | ongoing events should take place and | be listed as ongoing in the safety table. | In addition, the PI will ensure that the | Financial Disclosure Statements will be | completed by the PI and the Sub- | Investigator upon entry into the study | and as any changes that affect their | financial disclosure status occur during |
| Item | | | | | | | | | | | Investigator | Obligations | (Financial<br>Disclosure) | | | |
| Page | | | | | | | | | | | 49 | | | | | |
| Version Page | | | | | | | | | | | | | | | | |

| Study Protocol—Device | % smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | |

| Reason | | | egular Clarification implemented | | source remospective study | | | | | subject, Clarification implemented | | ive study. | | nination of | g. safety | end of the | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| New | | | The Sponsor will designate a monitor to conduct regular | monitoring visits. The purpose of these visits are to ensure | that data is accurate, complete and verifiable from source | documents. | | | | The end of study is defined as the date of the last subject, | last visit (LSLV). No additional care for subjects will be | provided under the protocol as this is a retrospective study. | | Should circumstances arise which require the termination of | the entire study prior to its planned completion (e.g. safety | concerns) or circumstances arise which mean the end of the | |
| Original | the course of the study and up to one | year after study completion. | The Sponsor will designate a monitor | to conduct regular monitoring visits. | The purpose of these visits are to | ensure the wellbeing of the subjects | are protected and that data is accurate, | complete and verifiable from source | documents. | The end of study is defined as the date | of the last subject, last visit (LSLV). No | additional care for subjects will be | provided under the protocol will be | provided once their participation in the | study has ended. | Should circumstances arise which | : : |
| Item | | | Sponsor and | Monitor | Opligations | | | | | End of Study | | | | | | | |
| Version | | | | | | | | | | | | | | | | | |

| Study Protocol—Device | > smith&nephew |
|---|---|
| DMCF Study on DEFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Page: 17</b> of <b>63</b> |

| Reason | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| New | Investigator, non-compliance), then this will be undertaken | according to the SOPs of the Sponsor. | | | | | | | | | | | | | |
| Original | study prior to its planned completion | (e.g. safety concerns) or circumstances | arise which mean the end of the | participation of an individual site (e.g. | departure of Investigator, non- | compliance), then this will be | undertaken according to the SOPs of | the Sponsor. Al <del>l reasonable efforts</del> | should be made to retain the subjects | for the 12-month post-operative follow- | up of this study. A study termination | CRF needs to be completed for any | subject that does not complete the | study, to document the reason for | termination. |
| ltem | | | | | | | | | | | | | | | |
| Page | | | | | | | | | | | | | | | |
| Version | | | | | | | | | | | | | | | |

| Study Protocol—Device | > smith&nephew |
|---|---|
| PMCF Study on PFFK Suture Anchors for Hin | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Page: 18</b> of <b>63</b> |

| Reason | Clarification implemented as it is applicable for a retrospective study. |
|---|---|
| New | If a subject has bilateral implants and has a revision, both implants will continue to be followed per the protocol visit schedule. |
| Original | Revision of the If a subject has bilateral implants and Study Device has a revision, the subject will be maintained in the study and both implants will continue to be followed per the protocol visit schedule |
| ltem | Revision of the<br>Study Device |
| Page | 50 |
| Version Page | |

# 3. SPONSOR APPROVAL

| | Job title | DocuSign Stamp |
|---|---|---|
| Sr. Vice President, Chief<br>Medical Officer, Global<br>R&D | Weymann, Andy | DocuSigned by: Signer Name: Andy Weymann Signing Reason: I approve this document Signing Time: 08-Apr-2019 16:52 BST 675C45EC25704A5FB20A08674419D6D8 |
| Head of Global Clinical<br>Strategy | Hanson, Beate | DocuSigned by: Brate Hanson Signer Name: Beate Hanson Signing Reason: I approve this document Signing Time: 08-Apr-2019 16:06 BST A491AB16277146CA9C8B8366F1B6BEA5 |
| Head of Global<br>Biostatistics and Data<br>Management | Rossington, Alan | DocuSigned by: Compared the content of the conte |
| Medical Affairs<br>Representative | Orlandini, Luca | DocuSigned by: Luca Orlandini Signing Reason: I approve this document Signing Time: 05-Apr-2019 17:26 BST FC872951AC1C4261B85EC7A7CD09ACDC |

# ****

# 4. SYNOPSIS

| Title of Study: | PMCF Study on PEEK Sutur | re Anchors for Hip Indications |
|---|---|---|
| Study Design: | Multi-center, retrospective | case series. |
| Study Type: | Post-market Clinical Follow | v-up |
| | PEEK Suture Anchors for Hi<br>*Part numbers as of Septer | Part numbers as of September 2018 |
| Study Products: | Suture Anchor | |
| | SpeedLock Hip Suture<br>Anchor | nchor |
| Intended Use: | The PEEK anchors are intellibring following hip capsule re | nded to be used for soft tissue to bone fixation in the epair. |
| Study Purpose: | Assess safety and perform to address clinical data ga | nance post-market of the PEEK suture anchor devices ps for MDR. |
| Primary Outcome: | Evidence of safety and per hip. | formance of the PEEK suture anchor devices in the |
| Statistical Rationale: | recruitment, enrolment and powered for any statistical | udy is determined based on the feasibility of d follow-up considerations. The study is therefore not hypothesis testing but will be able to estimate a with a 95% confidence interval (CI) of 80% to 100%. |
| | Minimum number of subje | cts, n=40 |
| | Maximum number of subje | ects, n=240 |
| | Enrollment distribution: | |
| Sample Size: | | a maximum of 40 subjects per anchor configuration 0 subjects will be enrolled for any anchor type. |

# ****

| | PEEK Anchor | Minimum<br>Number of<br>Subjects/Site | Maximum<br>Number of<br>Subjects/Site | Maximum Number of Subjects for the Study |
|---|---|---|---|---|
| | Bioraptor Knotless<br>Suture Anchor | 20 subjects per<br>site | 40 subjects per site | 120 subjects |
| | SpeedLock Hip | 20 subjects per<br>site | 40subjects per site | 120 subjects |
| | Total | 40 subjects | 80 subjects | 240 subjects |
| Number of Study<br>Sites: | Up to 6 sites | | | |
| Targeted Global<br>Regions: | USA | | | |
| Inclusion Criteria: | <ol> <li>Subjects who have undergone hip joint repair using the study devices.</li> <li>Subjects aged 18 years and older at the time of surgery.</li> <li>Subjects must have had a visit to their provider between 6 and 15 months post-operative.</li> </ol> | | | |
| Exclusion Criteria: | Subject is entered study or has prior to surge | <ol> <li>Subjects who are &lt; 12 months post-operative.</li> <li>Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 30 days prior to surgery.</li> </ol> | | |
| Study Duration: | Twelve month follow- | up | | |
| Primary Endpoint: | Clinical success rate ( | (%) at 6 months post- | operative based on s | standard of care |
| Secondary<br>Endpoint: | Clinical success rate (%) at 12 months post-operative based on standard of care | | | |
| Exploratory<br>Outcomes: | chart as standard of c | Surgeon Reported Outcomes based on data collected on the subject's medical chart as standard of care at study sites. These may include but not restricted to | | |
| | the following: | | | |

# ****

| Study Protocol—Device | *smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

| | Range of Motion (ROM) |
|---|---|
| | Flexion |
| | Extension |
| | <ul> <li>Abduction</li> </ul> |
| | <ul> <li>Adduction</li> </ul> |
| | External/Internal Rotation |
| | Pain assessed by VAS |
| | <ul> <li>All AEs, SAEs and complications including intra-operative adverse<br/>events and complications.</li> </ul> |
| Safety Endpoints: | Device related intervention |
| | Device deficiency |

# ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| , | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

# 5. SCHEDULE OF EVENTS

# **Table 1: Schedule of Events**

| Schedule of Events | Chart Review | |
|---|---|---|
| | 182 days post-op | 365 days post-op |
| | 6M (±91 Days) | 12M (± 91 Days ) |
| Informed Consent | X NA if waiver of consent granted by | |
| | IRB | |
| Inclusion/Exclusion | X | |
| Demographics/Medical<br>History | X | |
| VAS, ROM | X | Х |
| Operative Data Collection | X | |
| Implant Status and / or Disposition | X | X |
| Concomitant Medications or Therapies <sup>1</sup> | X | X |
| AE, SAE and DevD<br>Assessment | Х | X |
| End of Study | | X <sup>2</sup> |

# ****

<sup>&</sup>lt;sup>1</sup> Any concomitant medications associated with an AE, SA(D)E will be recorded.

<sup>&</sup>lt;sup>2</sup> End of Study CRF can be completed at 6 months if the subject did not have a 12-month visit.

# Study Protocol—Device

# PMCF Study on PEEK Suture Anchors for Hip Indications



Number: 2018.14.SMD.PEEK.RET.HIP


# 6. TABLE OF CONTENTS

| 1. | Signatures | 2 |
|------|-----------------------------------------------|----|
| 1.1 | Protocol Signature Page | 2 |
| 2. | Revision History, Ownership, and Approvals: | 3 |
| 2.1 | Revision History | 3 |
| 3. | Sponsor Approval | 19 |
| 4. | Synopsis | 20 |
| 5. | Schedule of events | 23 |
| 6. | Table of Contents | 24 |
| 7. | List of Abbreviations | 27 |
| 8. | Introduction | 29 |
| 8.1 | Study Purpose | 30 |
| 8.2 | Safety Considerations | 30 |
| 9. | Objective | 30 |
| 9.1 | Primary Objective | 30 |
| 10. | Study Product(s) | 31 |
| 10.1 | BIORAPTOR <sup>®</sup> Knotless Suture Anchor | 31 |
| 10.2 | SpeedLock Hip Suture Anchor | 32 |
| 10.3 | Indications | 32 |
| 10.4 | Product Use | 33 |
| 11. | Subject Enrollment and Withdrawal | 33 |
| 11.1 | Subject Population | 33 |
| 11.2 | Inclusion Criteria | 33 |
| 11.3 | Exclusion Criteria | 34 |
| 11.4 | Screening | 34 |
| 11.5 | Informed Consent | 34 |

# ****

# Study Protocol—Device

# PMCF Study on PEEK Suture Anchors for Hip Indications



Number: 2018.14.SMD.PEEK.RET.HIP


| 11. | 6 | Enrollment | . 35 |
|---|---|---|---|
| 11. | 7 | Lost to Follow-Up | . 35 |
| 11. | 8 | Withdrawal | . 35 |
| 12. | Stud | dy Design | . 36 |
| 12. | 1 | Study Design | . 36 |
| 12. | 2 | Allocation and Blinding | . 36 |
| 12. | 3 | Study Endpoints | . 37 |
| 13. | Stud | dy Procedures | . 38 |
| 13. | 1 | 6 months Post-Op Chart Review | . 38 |
| 13. | 2 | 12 months post-op Chart Review | . 39 |
| 13. | 3 | Concomitant Medications and Therapies | . 39 |
| 14. | Stat | istical Design | . 39 |
| 14. | 1 | General | . 39 |
| 14. | 2 | Analysis Populations | . 40 |
| 14. | 3 | Efficacy Analysis | . 40 |
| 14. | 4 | Safety Analyses | 41 |
| 14. | 5 | OTHER ENDPOINT Analyses | . 42 |
| 15. | San | nple Size Justification | . 42 |
| 16. | Adv | erse Events and Device Deficiencies | . 43 |
| 16. | 1 | Definitions | . 43 |
| 16. | 2 | Reporting Procedures | . 47 |
| 17. | Inve | estigator Obligations | . 49 |
| 18. | Sponsor and Monitor Responsibilities | | |
| 19. | Prot | ocol Amendments | . 49 |
| 20. | Con | fidentiality of the Study | . 49 |
| 21. | Stat | ements of Compliance | . 49 |

# ****

End of Study......50

| 23. | Revision of the Study Device | 50 |
|-------|---------------------------------------------------|----|
| 24. | Publication Policy | 51 |
| 24 | 4.1 Publication of Study Data | 51 |
| 24 | 4.2 Data Sharing | 51 |
| 25. | References | 52 |
| 26. | Appendices | 53 |
| 26 | 5.1 Principal Investigator Obligations (ISO14155) | 53 |
| | TABLES | |
| Table | e 1: Schedule of Events | 23 |
| Table | e 2: Instructions for Use Reference Numbers | 30 |
| Table | e 3: Part Numbers | 32 |
| Table | e 4: Enrollment | 36 |
| Table | e 5: Categories of Adverse Events | 44 |
| | FIGURES | |

# ****

This document contains information that is confidential and proprietary to Smith & Nephew PLC and Smith & Nephew, Inc. and is intended for use only by Smith & Nephew and its manufacturer. It shall not be reproduced or copied in whole or in part, nor shall the contents be disclosed by any means without prior written permission from Smith & Nephew, nor shall anyone make any use of it that is contrary to the expressed or implied wishes of Smith & Nephew.

22.

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| Indications | <b>Version:</b> 2.0, 03 April 2019 |

# 7. LIST OF ABBREVIATIONS

| Abbreviation | Term |
|--------------|----------------------------------------------------|
| ABHI | Association of British Healthcare Industries |
| ABS | Acrylonitrile Butadiene Styrene |
| ADE | Adverse Device Effect(s) |
| AE | Adverse Event(s) |
| ASADE | Anticipated Serious Adverse Device Effect |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval |
| CRF | Case Report Form(s) |
| CSR | Clinical Study Report |
| CTA | Clinical Trial Agreement |
| CV | Curriculum Vitae |
| DevD | Device Deficiency(ies) |
| GCP | Good Clinical Practice |
| HHS | Health and Human Services |
| ICH | International Conference on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | International Ethics Committee |
| IFU | Instructions for Use |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| ISO | International Organization for Standardization |
| LSLV | Last subject, last visit |

# ****

| Abbreviation | Term |
|--------------|------------------------------------------------|
| MDR | Medical Device Regulation |
| N (or n) | Total Sample Size (or subgroup sample size) |
| NA or N/A | Not Applicable |
| PEEK / PK | Polyetheretherketone |
| PI | Principal Investigator |
| PMCF | Post-market Clinical Follow-up |
| PP | Per-protocol Population |
| ROM | Range of Motion |
| S&N | Smith & Nephew Inc. |
| SADE | Serious Adverse Device Effect(s) |
| SAE | Serious Adverse Event(s) |
| SAF | Safety Population |
| SAP | Statistical Analysis Plan |
| USADE | Unanticipated Serious Adverse Device Effect(s) |
| VAS | Visual Analogue Scale |

# ****

# 8. INTRODUCTION

Suture anchors are small fixation devices used in surgical procedures for attaching or reattaching tendons and ligaments to bone. The size and type of anchor used depends on the patient's bone density and the procedure performed.

Suture anchors are made of three components: the anchor which is inserted into the bone; the eyelet – which is a hole or a loop in the anchor that the suture passes through to link the anchor to the suture; and the suture – which is attached to the anchor through the eyelet of the anchor. An anchor- receiving hole is first drilled in the bone at the desired point of tissue reattachment. A suture anchor is deployed in the hole using an appropriate installation tool. This effectively locks the suture to the bone, with the free end(s) of the suture extending out the bone. Soft tissue is then moved into position over the hole containing the deployed suture anchor. As this is done, the free end(s) of the suture is (are) passed through or around the soft tissue so that the free end(s) of the suture reside(s) on the far (i.e., non-bone) side of the soft tissue. The suture is now used to tie the soft tissue securely to the bone.

Smith & Nephew offers a variety of suture anchors including several polyetheretherketone (PEEK) suture anchors soft tissue to bone repair. The PEEK devices included in study are all single use, sterile devices comprised of machined component anchor bodies that are manufactured from PEEK-OPTIMA Polymer (LT1). This material meets ISO 10993 biocompatibility requirements for implant devices, bone/tissue contact and permanent contact. The anchor tips are molded components which are also manufactured from PEEK-OPTIMA Polymer (LT3). PEEK-OPTIMA polymers provide an ideal combination of strength, biocompatibility, reviseability and inherent radiolucent characteristics. Smith & Nephew also provides a variety of reusable and disposable

### ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| • | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

instrumentation used in conjunction with the suture anchors including awls, dilators, drills, guides, obturators and wires.

# **8.1 STUDY PURPOSE**

The purpose of this study is to conduct post-market clinical follow-up regarding the safety and performance of the PEEK anchors as required per MDR.

### **8.2 SAFETY CONSIDERATIONS**

Refer to the IFUs.

# **Table 2: Instructions for Use Reference Numbers**

Instructions for use document numbers have been provided as a reference but may not have been the version used at the time of surgery.

| PEEK Suture Anchor | IFU |
|----------------------------------|-----------------------------|
| Bioraptor Knotless Suture Anchor | 10600479 2/17, Rev E |
| SpeedLock Hip Suture Anchor | P/N 62513 March 2017, Rev B |

### 9. OBJECTIVE

#### 9.1 PRIMARY OBJECTIVE

The primary objective of this study is to assess safety and performance post-market of the PEEK anchor devices in the hip.

# ****

# 10. STUDY PRODUCT(S)

# 10.1 BIORAPTOR° KNOTLESS SUTURE ANCHOR



The BIORAPTOR° Knotless Suture Anchor is a single use, sterile, tap-in anchor that is manufactured from PEEK-OPTIMA® from Invibio®. The anchor is pre-assembled on an inserter comprised of a stainless steel shaft and an ABS and polycarbonate handle. The anchor is sized appropriately to facilitate both hip and shoulder procedures. The design consists of an outer anchor body and an inner shaft plug. The ribbed anchor, loaded with suture tails, is tapped into a pre-drilled prepared hole. The surgeon is now able to reapproximate the tissue to the appropriate tension and then use the torque-limiting knob on the insertion device that moves the inner plug down to lock the plug and achieve a secure fixation.

### ****

### 10.2 SPEEDLOCK HIP SUTURE ANCHOR



The SpeedLock Knotless Fixation Device is an implant that facilitates the attachment of tissue to bone. The SpeedLock system consists of a fixation device pre-loaded with a suture snare in an inserter handle. The SpeedLock implant is a knotless fixation device, in other words surgical knots are not necessary for fixation of suture to tissue.

### 10.3 INDICATIONS

The Smith & Nephew PEEK anchors are intended to be used for soft tissue to bone fixation in the hip following hip capsule repair.

**Table 3: Part Numbers** 

Peek Suture Anchors for the Hip

\*Part numbers as of September 2018

| Bioraptor Knotless Suture Anchor | 72202397 |
|----------------------------------|----------|
| SpeedLock Hip Suture Anchor | OM-7500 |

### ****

# **10.4 PRODUCT USE**

All study related procedures using the PEEK suture anchors in the hip have been performed according to the recommended surgical technique described in the labelling and the instructions for use.

### 11. SUBJECT ENROLLMENT AND WITHDRAWAL

Investigators will screen all subjects that have undergone usage of the PEEK suture anchors in the hip using only the existing information in the medical records.

Investigators will conduct a chart review after IRB approval has been granted. All subjects whose chart undergoes the screening process will be documented on a Screening and Enrollment Log, with the reason for exclusion noted, if applicable. The Investigator or designee must notify the Sponsor upon subject enrollment.

# 11.1 SUBJECT POPULATION

To minimize the potential for selection bias, Investigators will screen and subsequently enroll subjects (after fulfilling all inclusion and exclusion criteria) on whom PEEK suture anchors in the hip were implanted. Enrollment will be in sequential order based on the date of their surgical procedure with the investigational device, i.e. time of surgery to present day.

# 11.2 INCLUSION CRITERIA

# Subjects will be considered qualified for enrollment if they meet the following criteria:

- 1. Subjects who have undergone hip joint repair using the study devices.
- 2. Subjects aged 18 years and older at the time of surgery.

### ****

| Study Protocol—Device | *smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| • | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

3. Subjects must have had a visit to their provider between 3 and 15 months post-operative.

# 11.3 EXCLUSION CRITERIA

Any one (1) of the following criteria will disqualify a potential subject from participation in the study:

- 1. Subjects who are < 12 months post-operative.
- 2. Subject is entered in another investigational drug, biologic, or device study or has been treated with an investigational product within 30 days prior to surgery.
- 3. Subject had off-label use of the PEEK suture anchor during surgery.

#### 11.4 SCREENING

Participating study sites are required to document all screened subjects considered for inclusion in this study. If a subject is excluded from the study, the reasons for exclusion will be documented in the subject's source documents and noted on the Screening and Enrollment Log.

### 11.5 INFORMED CONSENT

For adults and children, a waiver or alteration of the requirements for obtaining informed consent can occur under any of the following three provisions set forth by HHS:

Research in general: an IRB may waive or alter the requirement of informed consent under <u>45</u> <u>CFR 46.116(d)</u>, provided that the IRB finds and documents that all of the following four conditions are met: [3]

- 1. the research involves no more than minimal risk to the participants;
- 2. the waiver or alteration will not adversely affect the rights and welfare of the participants;

#### ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| , | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

- 3. the research could not practicably be carried out without the waiver or alteration; and
- 4. whenever appropriate, the participants will be provided with additional pertinent information after participation.

#### 11.6 ENROLLMENT

Enrollment in this study shall occur when subjects have meet inclusion criteria and none of the exclusion criteria. When a subject is enrolled for the left hip as well as the right hip, only one subject ID will be allocated.

#### 11.7 LOST TO FOLLOW-UP

Not applicable.

### 11.8 WITHDRAWAL

# 11.8.1 Withdrawal from the Study

The Investigator may withdraw subjects from the study for many reasons, including but not limited to the following:

- At the discretion of the Investigator.
- If the Investigator or the Sponsor stops the study for any reason and decides to withdraw subject(s) from the study.

For each case, information will be documented in the source document and the Case Report Form (CRF), detailing circumstances leading to the withdrawal.

Subjects who are withdrawn will not be re-entered into the study at a later date. Data collected up to the point of withdrawal may be used but no additional data for that subject may be collected.

### ****

### 12. STUDY DESIGN

### 12.1 STUDY DESIGN

This is a retrospective, open-label, multi-center study to collect clinical data that will evaluate post-market safety and performance of the PEEK suture anchors in the hip. A minimum of 40 subjects and a maximum of 240 subjects in the United States who underwent surgery in the hip using the Smith & Nephew PEEK suture anchors are planned to be enrolled into the study after the fulfilment of all inclusion and exclusion criteria. Up to three sites will enroll a minimum of 20 subjects and a maximum of 40 subjects per anchor configuration; therefore, not more than 120 subjects will be enrolled for any anchor type.

Data obtained from enrolled eligible subjects will subsequently be recorded on case report forms.

Table 4: Enrollment

| PEEK Anchor | Minimum Number of<br>Subjects/Site | Maximum Number of Subjects/Site | Maximum Number of<br>Subjects for the Study |
|---|---|---|---|
| Bioraptor Knotless<br>Suture Anchor | 20 subjects per site | 40 per site | 120 subjects |
| SpeedLock Hip | 20 subjects per site | 40 per site | 120 subjects |
| Total | 40 subjects | 80 subjects | 240 subjects |

# 12.2 ALLOCATION AND BLINDING

This study is not randomized or blinded.

### ****
| Study Protocol—Device | smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

## 12.3 STUDY ENDPOINTS

# 12.3.1 Primary Endpoint

The primary endpoint will be clinical success rate (%) at 6 months post-operative based on standard of care. Clinical success is defined as hip repairs without signs of device failure and/or re-intervention as assessed by the surgeon.

# 12.3.2 Secondary Endpoints

The secondary endpoint will be clinical success rate (%) at 12 months post-operative based on standard of care. Clinical success has previously been defined. It is expected that per physician's standard of care, 12 month clinical data will be consistently be available.

# 12.3.3 Safety Endpoints

Safety endpoints will include but not restricted to the following events:

- All adverse events, SAEs and complications occurring from the time of enrollment until study termination or study completion including intra-operative adverse events and complications.
- Device related intervention.
- Device deficiency.

# 12.3.4 Other Endpoints

Surgeon Reported Outcomes would constitute other endpoints and may include but not restricted to the following:

- Range of Motion (ROM)
  - Flexion
  - Extension

## ****

| Study Protocol—Device | smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

- Abduction
- Adduction
- External/Internal Rotation
- Pain assessed by VAS

# 13. STUDY PROCEDURES

# 13.1 6 MONTHS POST-OP CHART REVIEW

NOTE: Any subject, who meets the inclusion/exclusion criteria, will be assigned a subject number.

- 1. Subject should undergo the informed consent process and sign the informed consent *only* if a waiver of consent has not been approved by the IRB.
- 2. Screen the subject's chart for protocol inclusion/exclusion criteria.
- 3. Obtain demographic information and a medical history.
- 4. VAS, ROM.
- 5. Operative Data Collection review operative case notes.
- 6. Implant Status / Disposition.
- 7. Document concomitant medications and/or therapies associated with an AE, SA(D)E
- 8. Review the subject's chart for AEs, SAEs and Device Deficiencies, including interoperative. AEs, SAEs and DevDs should be documented from the time of surgery through the study duration.

## ****

## 13.2 12 MONTHS POST-OP CHART REVIEW

- 1. VAS, ROM
- 2. Implant Status/Disposition
- 3. Document concomitant medications and/or therapies associated with an AE, SA(D)E
- Review the subject's chart for AEs, SAEs and Device Deficiencies including inter-operative.
   AEs, SAEs and DevDs should be documented from the time of surgery through the study duration.
- 5. Complete the End of Study CRF.

# 13.3 CONCOMITANT MEDICATIONS AND THERAPIES

Any concomitant medications associated with an AE, SAE or SADE will be recorded. Concomitant medications will be recorded from the time of surgery through 12 months. If the subject's final visit occurred at 6 months, concomitant medications will be collect through 6 months.

# 14. STATISTICAL DESIGN

A Statistical Analysis Plan (SAP) will be written and finalized prior to database lock. The analyses specified in the protocol will be a microcosm of the detailed analyses to be contained in the SAP. If there are changes to or additional analyses required to the analysis described below, it will be described in the SAP and the Clinical Study Report (CSR).

# 14.1 GENERAL

Smith & Nephew's Global Biostatistics group or designee will conduct the statistical analysis for this study. Unless otherwise stated, all significance tests will be two-sided, performed at the 5%

## ****

| Study Protocol—Device | smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

significance level. Resulting p-values will be provided and 95% two-sided confidence intervals will be generated where appropriate.

Where data summaries are specified, categorical and ordinal variables will be summarized with frequencies and percentages. Continuous variables will be summarized with the following summary statistics: number of observations, mean, median, standard deviation, minimum and maximum values. All analyses will be performed in SAS version 9.3 (or later).

# 14.2 ANALYSIS POPULATIONS

The following analysis populations will be used for this study:

- Safety Population (SAF): This includes all subjects who enroll in the study who had previously undergone hip repair using PEEK suture anchors, i.e. subjects who would provide retrospective data.
- **Per-Protocol Population (PP):** This includes all subjects in the Safety Population, who have no significant protocol deviations and who meet all the inclusion/exclusion criteria.

#### 14.3 EFFICACY ANALYSIS

# 14.3.1 Analysis of Primary Endpoint

The rate (%) of clinical success of all the PEEK suture anchor devices combined at 6 months post-operative will be summarized as a frequency and percentage. A 95% two-sided exact CI for a single proportion will be presented using Clopper-Pearson's method [1]. The same type analysis would be carried out for each of the 2 different PEEK suture anchors used in the study. These

## ****

| Study Protocol—Device | smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

analyses will be carried out using the per protocol population as the primary analysis population with the safety population used for sensitivity analysis.

# 14.3.2 Analysis of Secondary Endpoints

The analysis of the following secondary endpoint will be carried out using the safety population.

The rate (%) of clinical success of all the PEEK suture anchors combined at 12 months post-operative will be summarized as described for the analysis of the primary endpoint. This analysis will also be repeated for each of the 2 different types of PEEK suture anchors used in the study.

## 14.4 SAFETY ANALYSES

- All safety endpoints will be summarized using the safety population. The incidence of events encountered on study will be summarized using frequencies and percentages. An overall AE table will be summarized using the overall incidence according to subjects with at least one AE; subjects with at least one AE by worst severity (mild, moderate, or severe); subjects with at least one AE by worst outcome; subjects with one AE that led to study discontinuation; subjects with at least one AE by relatedness to investigational device; SAEs; ADEs; ASADEs; USADEs and SADEs as applicable. A cumulative summary by the number of events encountered within each classification will also be summarized. The incidence of subjects reporting device deficiencies will additionally be summarized.
- Each of the AE classifications will further be summarized by event using the frequencies
   (n) and percentages (%) of subjects with each event as well as the ccumulative events/episodes per event.
- A listing of concomitant medications will be provided by subject.

#### ****

| Study Protocol—Device | smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

Additional summaries of safety endpoints, if applicable, will be described in the SAP.

# 14.5 OTHER ENDPOINT ANALYSES

- The analyses of other endpoints will be carried out using the safety population. Overall, device-related failure and device-related re-intervention encountered on-study will be summarized independently as frequencies and percentages. A 95% two-sided exact CI for a single proportion will be presented for each proportion using Clopper-Pearson's method (1934).
- The derivation of surgeon reported outcomes used in summarizing this data for the study will be described in the SAP and will be summarized as appropriate using descriptive summary characteristics for continuous or categorical endpoints at 6 months and 12 months

# 13.6 Interim Analyses

Not applicable

## 15. SAMPLE SIZE JUSTIFICATION

This study is precision-based, as a result, the sample size is not based on statistical power calculations.

The sample size for this study is determined based on the feasibility of recruitment, enrollment and follow-up considerations. The study is therefore not powered for any statistical hypothesis testing but will be able to estimate a clinical success rate of 91% with a 95% confidence interval (CI) of 80% to 100%.

#### ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

With an assumption of a 91% clinical success rate to be obtained in each of the PEEK anchor sutures and a corresponding 95% CI between 80% and 100%, enrolling between 20 and 120 subjects for each PEEK anchor suture's precision analysis will provide between 15.2% to 95% probability. Thus, an overall minimum of 40 and maximum of 240 subjects who had previously undergone surgery of the hip using PEEK anchor sutures will be enrolled into the study. Additionally, a minimum of 20 subjects will be enrolled at any investigational site.

# 16. ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### **16.1 DEFINITIONS**

The categories of adverse events are shown in Table 4. The definitions for each of these categories are given in the subsequent sections (see reference within the table). All adverse events will be captured from the time of surgery through the 12-month follow-up visit.

[Intentionally left blank]

## ****

| Study Protocol—Device | *smith&nephew |
|-----------------------|----------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

**Table 5: Categories of Adverse Events** 

| | NOT DEVICE-<br>RELATED | DEVICE- OR PROCEDURE-RELATED | |
|---|---|---|---|
| NON-<br>SERIOUS | ADVERSE EVENT<br>(AE) | Adverse Device Effect (ADE) | |
| | SERIOUS ADVERSE | SERIOUS ADVERSE DEVICE EFFECT (SADE) | |
| SERIOUS | EVENT (SAE) | ANTICIPATED | UNANTICIPATED |
| | (SAE) | ANTICIPATED SERIOUS<br>ADVERSE DEVICE EFFECT<br>(ASADE) | UNANTICIPATED SERIOUS<br>ADVERSE DEVICE EFFECT<br>(USADE) |

# 16.1.1 Adverse Event

An <u>Adverse Event (AE)</u> is any untoward medical occurrence temporally associated with the use of an IP/Ancillary Product, whether or not considered causally related to that IP/Ancillary Product. AE is used both to refer to AE which are non-serious non-IP or procedure-related and as an umbrella term referring to adverse events of all classifications.

An AE can be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease. For reporting purposes, emphasis is placed first and foremost on whether or not the event constitutes an <u>untoward medical occurrence</u>.

## 16.1.2 Adverse Device Effect

An <u>Adverse Device Effect (ADE)</u> is an adverse event that, in the opinion of the investigator, is related to the IP or the procedure.

## ****

| Study Protocol—Device | *smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

Not Related - An AE is considered to be not related to the use of an IP or the procedure when the effect is DEFINITELY UNRELATED or UNLIKELY to have any relationship to the use of the IP or the procedure.

Related – An AE is considered to be related to the use of an IP or the procedure when there is a POSSIBLE, PROBABLE, or DEFINITE relationship between the AE and the use of the IP or the procedure.

# 16.1.3 Serious Adverse Events and Serious Adverse Device Effects

An AE or ADE is considered a **Serious** Adverse Event (SAE) or **Serious** Adverse Device Effects (SADE) if, in the view of either the Investigator or the Sponsor, it:

- Results in death.
- Is life-threatening (*NOTE*: The term "life-threatening" in the definition of "serious" refers to an event/reaction in which the subject was at risk of death at the time of the event/reaction; it does not refer to an event/ reaction which hypothetically might have caused death if it were more severe).
- Requires in subject hospitalization or results in prolongation of existing hospitalization.
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- Is a congenital anomaly/birth defect.
- Is a medically important event or reaction.

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious such as important medical events that might not be immediately life

## ****

#### 

threatening or result in death or hospitalization but might jeopardize the subject or might require intervention to prevent one of the other outcomes listed in the definition above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

# 16.1.4 Anticipated/Unanticipated Serious Adverse Device Effect

An Unanticipated Serious Adverse Device Effect (USADE) is a serious ADE that meets any of the above definitions but is also considered, by the Investigator, to be caused by or related to the IP, not previously identified in nature, severity or degree in the IFU.

An Anticipated Serious Adverse Device Effect (ASADE) is a serious ADE that does not meet the criteria for a USADE.

# 16.1.5 Severity

The severity of every AE will be assessed by the PI or medically qualified site staff to whom the responsibility has been delegated and documented on the delegation of authority log. AE should be classified as mild, moderate, or severe, regardless of whether or not the AE are considered to be serious or non-serious. The classification should be based on the following definitions:

 An event is mild if the subject is aware of, but can easily tolerate the sign or symptom.

**Moderate** - An event is moderate if the sign or symptom results in discomfort significant enough to cause interference with the subject's usual activities.

## ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

Severe - An event is severe if the sign or symptom is incapacitating and results in the subject's inability to work or engage in their usual activities.

# 16.1.6 Device Deficiency

A Device Deficiency (DevD) is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. DevD includes malfunctions, use errors and inadequate labelling.

## **16.2 REPORTING PROCEDURES**

AE of any kind and DevD will be recorded in the applicable CRF and source notes. The Investigator will evaluate all AE for relationship to the device and procedure, if applicable, seriousness, and severity. ADE, SAE, and DevD will be entered into the CRF and reported to the Sponsor within 24 hours of the investigator being informed about the event (Figure 1). Applicable to the retrospective study design, 24 hour reporting begins at the time the Investigator was informed of the event under the auspice of the clinical study. For ADE and DevD, details of the product/procedure related to the event will be included and where applicable and available, pictures taken of the device. If available the deficient product should be retained for return to S&N unless it is contaminated (e.g. used dressings must not be retained).

All SAE and ADE will be reviewed by a medically qualified person appointed by the Sponsor to determine which, if any, meet criteria for expedited reporting to the regulatory authorities. The investigator will inform the IRB/IEC of adverse events according to the IRB/IEC requirements. Depending on the nature of the adverse event, S&N may request copies of the subject's medical records, imaging, operative notes, as well as results of any relevant laboratory tests performed or

## ****

| Study Protocol—Device | *smith&nephew |
|-----------------------|----------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

other documentation related to the AE. If the subject was hospitalized, a copy of the discharge summary may be requested by S&N and should be forwarded as soon as it becomes available. In certain cases, S&N also may request a letter from the Investigator that summarizes the events related to the case.

Figure 1: Evaluation and Reporting of AE and DevD



#### ****

| Study Protocol—Device | smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

Reference the ISF Sponsor Contact Information Sheet to report SAE, unanticipated ADE and SADE, anticipated SADE, and DevD.

## 17. INVESTIGATOR OBLIGATIONS

The Principal Investigator will comply with the commitments outlined in the Statement of Investigator, provided by the Sponsor, and with Good Clinical Practice (GCP), and all applicable regulatory requirements as outlined in Section 26.1 of this protocol.

# 18. SPONSOR AND MONITOR RESPONSIBILITIES

The Sponsor will designate a monitor to conduct regular monitoring visits. The purpose of these visits are to ensure that data is accurate, complete and verifiable from source documents.

## 19. PROTOCOL AMENDMENTS

Amendments should be made only in exceptional cases once the study has started. Protocol amendments must be approved by the protocol signatories prior to submission to the IRB. Protocol amendments need to be approved by the IRB and Regulatory Authority (ies), as applicable prior to implementation at the site.

#### 20. CONFIDENTIALITY OF THE STUDY

The confidentiality of this study and associated documents is governed by the terms of the Clinical Trial Agreement (CTA).

# 21. STATEMENTS OF COMPLIANCE

This clinical study will be performed in compliance with the ethical principles of the Declaration of Helsinki; ISO 14155: Clinical investigation of medical devices – Good Clinical Practice and ICH-E6.

## ****

Study Protocol—Device

PMCF Study on PEEK Suture Anchors for Hip

**Indications** 

smith&nephew

Number: 2018.14.SMD.PEEK.RET.HIP


This clinical study will not commence until the required approval/favorable opinion from the IRB or regulatory authority has been obtained. Any additional requirements imposed by the IRB or regulatory authority will be followed.

Public/Products Liability Insurance has been purchased by Smith & Nephew plc. Worldwide and incorporates coverage for personal injury in respect of clinical studies. The Sponsor agrees to operate in good faith and in accordance with ABHI (Association of British Healthcare Industries) guidelines regarding compensation for injury arising in the course of clinical studies.

# 22. END OF STUDY

The end of study is defined as the date of the last subject, last visit (LSLV). No additional care for subjects will be provided under the protocol, as this is a retrospective study.

Should circumstances arise which require the termination of the entire study prior to its planned completion (e.g. safety concerns) or circumstances arise which mean the end of the participation of an individual site (e.g. departure of Investigator, non-compliance), and then this will be undertaken according to the SOPs of the Sponsor.

# 23. REVISION OF THE STUDY DEVICE

If a subject has bilateral implants and has a revision, both implants will continue to be followed per the protocol visit schedule.

## ****

## 24. PUBLICATION POLICY

# **24.1 Publication of Study Data**

The preparation and submission for publication of manuscripts containing the study results shall be in accordance with a process determined by the Clinical Trial Agreements between the study Sponsor and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to the Health Insurance Portability and Accountability Act of 1996.

# **24.2 DATA SHARING**

Smith & Nephew is committed to upholding the highest ethical and legal standards involved in conducting clinical trials. Smith & Nephew therefore supports the data sharing requirements of The International Committee of Medical Journal Editors (ICMJE) published on the 6th June 2017 [2]. In accordance, Smith & Nephew will consider requests to share individual (de-identified) participant data that underlie the results of any interventional clinical trial, as presented from the 1st July 2018 within an ICMJE associated journal. Requests made by researchers who provide a methodologically sound proposal will be considered. Requests may include data that underlie results presented in text, tables, figures and appendices, together with data dictionaries. Availability of these data will begin 9 months and end 36 months after article publication. Data supplied may only be used by the researcher(s) named in the approved research proposal for the purposes of achieving the aims of the analyses specified therein. All proposals should be directed to datasharing.gcs@smith-nephew.com. To gain access, data requestors will need to sign a data access agreement.

## ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| • | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

# 25. REFERENCES

- 1. Clopper, CJ & Pearson ES. (1934) The use of confidence or fiducial limits illustrated in the case of the binomial. *Biometrika*, 26, 404–413.
- Taichman, DB, et al. Data Sharing Statements for Clinical Trials: A Requirement of the International Committee of Medical Journal Editors. Ann Intern Med. 2017. 6th June. doi:10.7326/M17-1028

# ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| • | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

## 26. APPENDICES

# **26.1 Principal Investigator Obligations (ISO14155)**

#### General:

a. The role of the PI is to implement and manage the day-to-day conduct of the clinical investigation as well as ensure data integrity and the rights, safety, and well-being of the subjects involved in the clinical investigation.

# 2. Qualification of the PI. The PI shall:

- a. be qualified by education, training, and experience to assume responsibility for the proper conduct of the clinical investigation in accordance with this International Standard; evidence of such qualifications of the PI and key members of the investigation site team shall be provided to the Sponsor through up-to-date Curriculum Vitae (CV) or other relevant documentation,
- b. be experienced in the field of application and trained in the use of the investigational device under consideration,
- c. disclose potential conflicts of interest, including financial, that interfere with the conduct of the clinical investigation or interpretation of results, and
- d. be knowledgeable with the method of obtaining informed consent.
- 3. Qualification of investigation site. The PI shall be able to demonstrate that the proposed investigation site:
  - has the required number of eligible subjects needed within the agreed recruitment period, and

## ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

b. has one or more qualified investigators, a qualified investigation site team and adequate facilities for the foreseen duration of the clinical investigation.

- 4. Communication with the IEC. The PI shall:
  - a. provide the Sponsor with copies of any clinical-investigation-related communications between the PI and the IEC,
  - b. comply with the requirements described in 4.5 of ISO 14155:
    - i. Submit to the IEC the following information, any amendments and any additional documentation required by the IEC: the Protocol; IB or equivalent; informed consent form and any other written information provided to subjects; procedures for recruiting subjects and advertising materials, if any; a copy of the CV of the PI(s) for with the IEC has oversight.
    - ii. Provide documentation of the IECs approval/favorable opinion, identifying the documents and amendments on which the opinion was based, to the Sponsor, prior to commencing the clinical investigation.
    - iii. Submit the following to the IEC if required by national regulations, the protocol or IEC, whichever is more stringent:
      - SAEs
      - Requests for deviations, and reports of deviations, if the deviation affects subject's rights, safety, and well-being, or the scientific integrity of the clinical investigation. Document and report to the Sponsor and IEC a report of deviations made to protect the rights, safety, and well-being of human subjects under emergency circumstances.
      - 3. Progress reports, including safety summary and deviations

## ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

- 4. Amendments to any documents already approved by the IEC.
- 5. If applicable, notifications of suspension or premature termination
- 6. If applicable, justification and request for resuming the clinical investigation after suspension.
- 7. Clinical investigation report or summary.
- iv. As a minimum, during the clinical investigation, the following information shall be obtained in writing from the IEC prior to implementation:
  - Approval/favorable opinion of amendments
  - Approval of the request for deviations that can affect the subject's rights, safety, and well-being or scientific integrity of the clinical investigation
  - 3. Approval for resumption of a suspended clinical investigation if applicable.
- obtain the written and dated approval/favorable opinion of the IEC for the clinical investigation before recruiting subjects and implementing all subsequent amendments, if required,
- d. promptly report any deviations from the protocol that affect the rights, safety or well-being of the subject or the scientific integrity of the clinical investigation, including those which occur under emergency circumstances, if required by the IEC, protocol or national regulations. In particular circumstances, the communication with the IEC can be performed by the Sponsor, partly or in full, in which case the Sponsor shall keep the Principal Investigator informed.
- 5. Informed consent process. The PI shall:
  - a. General:

#### 

- Informed consent shall be obtained in writing from the subject and the process shall be documented before any procedure specific to the clinical investigation is applied to the subject; except when special circumstances for emergency treatments apply (see below)
- ii. The informed consent form consists of an information form and informed consent signature form. These two forms can either be combined in one document or separated into two documents
- b. Process of obtaining informed consent. The general process for obtaining informed consent shall be documented in the protocol and shall comply with the following. These requirements also apply with respect to informed consent obtained from a subject's legally authorized representative:
  - i. Ensure that the PI or his/her authorized designee conducts the informed consent process
  - ii. Include all aspects of the clinical investigation that are relevant to the subject's decision to participate throughout the clinical investigation
  - iii. Avoid any coercion or undue improper influence on, or inducement of, the subject to participate
  - iv. Not waive or appear to waive the subject's legal rights
  - v. Use native non-technical language that is understandable to the subject
  - vi. Provide ample time for the subject to read and understand the informed consent form and to consider participation in the clinical investigation
  - vii. Include personally dated signatures and the PI or an authorized designee responsible for conducting the informed consent process

## ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

- viii. Show how informed consent will be obtained in special circumstances (see below) where the subject is unable to provide him or herself, and
- ix. Ensure important new information is provided to new and existing subjects throughout the clinical investigation.
- Special circumstances for informed consent (the following provisions are subject to national regulations):
  - i. Subject needing legally authorized representatives: the legally authorized representative may give informed consent only if a subject is unable to make the decision to participate in a clinical investigation (e.g. infant, child, or juvenile, seriously ill or unconscious subject, mentally ill person, mentally handicapped person). In such cases, the subject shall also be informed about the clinical investigation within his/her ability to understand.
  - ii. Subject unable to read or write: informed consent shall be obtained through a supervised oral process if a subject or legally authorized representative is unable to read or write. An independent witness shall be present throughout the process. The written informed consent form and any other information shall be read aloud and explained to the prospective subject or his/her legally authorized representative and, whenever possible, either shall sign and personally date the informed consent form. The witness also signs and personally dates the informed consent for attesting that the information was accurately explained and that the informed consent was freely given.
  - iii. Emergency treatments:

#### 

- For clinical investigations involving emergency treatments, when prior informed consent of the subject is not possible because of the subject's medical condition, the informed consent of the subject's legally authorized representative, if present, shall be requested.
- When it is not possible to obtain prior informed consent from the subject, and the subject's legally authorized representative, is not available, the subject may still be enrolled if a specific process has been described in the protocol.
- 3. Arrangements shall be made to inform the subject or legally authorized representative, as soon as possible, about the subject's inclusion in the clinical investigation and about all aspects of the clinical investigation.
- 4. The subject shall be asked to provide informed consent for continued participation as soon as his/her medical condition allows.
- d. The Principal Investigator may not enroll a subject without obtaining informed consent of the subject or his/her legally authorized representative only when the following conditions are fulfilled: the prospective subject fulfils the emergency conditions and is obviously in a life-threatening situation; no sufficient clinical benefits are anticipated from the currently available treatment; there is a fair possibility that the life-threatening risk to the prospective subject can be avoided if the investigational device is used; anticipated risks are outweighed by the potential benefits of applying the investigational device; the legally authorized representative cannot be promptly reached and informed.
- e. Information provided to the subject. All information pertinent to the clinical investigation, including at least the following, shall be provided in writing and in native, non-technical

## ****

#### 

language that is understandable to the subject (or the subject's legally authorized representative):

- i. Description and purpose
- ii. Potential benefits
- Risks and inconveniences or the subject and, when applicable, for any embryo, foetus or nursing infant
- iv. Alternative procedures
- v. Confidentiality
- vi. Compensation
- vii. Anticipated expenses, if any, to be borne by the subject for participating in the clinical investigation
- viii. Information on the role of Sponsor's representative in the clinical investigation
- ix. Contact persons
- x. Statement declaring that new findings or the reasons for any amendment to the protocol that affect the subject's continued participation shall be made available to the subject.
- xi. Statement indicating that, upon the subject's approval, the subject's personal physician will be informed of the subject's participation in the clinical investigation
- xii. Termination procedures
- f. Informed consent signature shall contain the following:
  - The voluntary agreement to participate in the clinical investigation and follow the investigator's instructions
  - ii. A statement declaring that refusal of participation incurs no penalty for the subject

## ****

| Study Protocol—Device | smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip | Number: 2018.14.SMD.PEEK.RET.HIP |
| , | <b>Version:</b> 2.0, 03 April 2019 |
| Indications | |

- iii. A statement declaring that discontinuation at any time incurs no penalty for the subject
- iv. A statement with regard to the possible consequences of withdrawal
- v. An acknowledgement of the information provided and confirmation that all the subject's questions were answered
- vi. A statement confirming that the subject or his/her legally authorized representative agrees to the use of the subject's relevant personal data for the purpose of the clinical investigation
- vii. A statement confirming that the subject or his/her legally authorized representative agrees that Sponsor's representatives, regulatory authorities and IEC representatives will be granted direct access to the subject's medical records.
- g. New information: if new information becomes available that can significantly affect a subject's future health and medical care, that information shall be provided to the subject(s) affected in written form. If relevant, all affected subjects shall be asked to confirm their continuing consent in writing.
- ensure compliance with the applicable regulatory requirements and ethical principles for the process of obtaining informed consent, and
- ensure and document appropriate training if an authorized designee is appointed to conduct the informed consent process.
- 6. Compliance with the protocol. The Principal Investigator shall:
  - a. indicate his/her acceptance of the protocol in writing,
  - b. conduct the clinical investigation in compliance with the protocol,

| Study Protocol—Device | > smith&nephew |
|-----------------------|------------------------------------|
| Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

- c. create and maintain source documents throughout the clinical investigation and make them available as requested during monitoring visits or audits,
- d. ensure that the investigational device is used solely by authorized users as specified in6.2, and in accordance with the protocol and instructions for use,
- e. propose to the Sponsor any appropriate modification(s) of the protocol or investigational device or of the use of the investigational device,
- f. refrain from implementing any modifications to the protocol without agreement from the Sponsor, IEC and regulatory authorities, if required,
- document and explain any deviation from the approved protocol that occurred during the course of the clinical investigation,
- h. ensure that an adequate investigation site team and facilities exist and are maintained and documented during the clinical investigation,
- ensure that maintenance and calibration of the equipment relevant for the assessment of the clinical investigation is appropriately performed and documented, where applicable,
- j. ensure the accuracy, completeness, legibility and timeliness of the data reported to the Sponsor in the CRF and in all required reports,
- k. maintain the device accountability records,
- l. allow and support the Sponsor to perform monitoring and auditing activities,
- m. be accessible to the monitor and respond to questions during monitoring visits,
- n. allow and support regulatory authorities and the IEC when performing auditing activities,
- ensure that all clinical-investigation-related records are retained as required taking measures to prevent accidental or premature destruction, and

| Study Protocol—Device | *smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

- p. review and sign the clinical investigation report, as applicable.
- 7. Medical care of subjects. The Principal Investigator shall
  - a. provide adequate medical care to a subject during and after a subject's participation in a clinical investigation in the case of adverse events,
  - b. inform the subject of the nature and possible cause of any adverse events experienced,
  - c. provide the subject with the necessary instructions on proper use, handling, storage, and return of the investigational device, when it is used or operated by the subject,
  - d. inform the subject of any new significant findings occurring during the clinical investigation, including the need for additional medical care that may be required,
  - e. provide the subject with well-defined procedures for possible emergency situations
    related to the clinical investigation, and make the necessary arrangements for
    emergency treatment, including decoding procedures for blinded/masked clinical
    investigations, as needed,
  - f. ensure that clinical records are clearly marked to indicate that the subject is enrolled in a particular clinical investigation,
  - g. if appropriate, subjects enrolled in the clinical investigation shall be provided with some means of showing their participation in the clinical investigation, together with identification and compliance information for concomitant treatment measures (contact address and telephone numbers shall be provided),
  - inform, with the subject's approval or when required by national regulations, the subject's personal physician about the subject's participation in the clinical investigation, and

| Study Protocol—Device | *smith&nephew |
|---|---|
| PMCF Study on PEEK Suture Anchors for Hip Indications | Number: 2018.14.SMD.PEEK.RET.HIP |

- make all reasonable efforts to ascertain the reason(s) for a subject's premature withdrawal from the clinical investigation while fully respecting the subject's rights.
- 8. Safety reporting. The Principal Investigator shall:
  - record every adverse event and observed device deficiency, together with an assessment,
  - report to the Sponsor, without unjustified delay, all serious adverse events and device deficiencies that could have led to a serious adverse device effect; this information shall be promptly followed by detailed written reports, as specified in the protocol,
  - c) report to the IEC serious adverse events and device deficiencies that could have led
    to a serious adverse device effect, if required by the national regulations or protocol or
    by the IEC,
  - d. report to regulatory authorities serious adverse events and device deficiencies that could have led to a serious adverse device effect, as required by the national regulations, and
  - e. supply the Sponsor, upon Sponsor's request, with any additional information related to the safety reporting of a particular event.